CLINICAL TRIAL: NCT02754687
Title: Single Dose, Dose-Ranging Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics Study of 11-β Methyl Nortestosterone Dodecylcarbonate (11β-MNTDC) in Healthy Men
Brief Title: Single Dose, Dose-Ranging Study of 11-β Methyl Nortestosterone Dodecylcarbonate (11β-MNTDC) in Healthy Men
Acronym: CCN014
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Washington (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCN014; HHSN275201200002I (Other Grant/Funding Number: NICHD Contract. This is not a grant but a contract.)
Record Dates: First submitted 2016-03-28; First posted 2016-04-28 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy Men; Male Contraception
Keywords: male contraception; healthy men; androgen; Nortestosterone; Dodecylcarbonate; 11-Beta; 11β; contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 11βmethyl nortestosterone dodecylcarbonate (Experimental): 11β-MNTDC in doses of 100 mg, 200 mg, 400 mg, and 800 mg
  Interventions: Drug: 11βmethyl nortestosterone dodecylcarbonate

INTERVENTIONS:
Drug: Placebo — Placebo with capsules that look like the 11β-MNTDC capsules but with no active ingredients
  Arms: Placebo
Drug: 11βmethyl nortestosterone dodecylcarbonate — Escalating doses of 100, 200, 400, and 800 mg 11β-MNTDC
  Other Names: 11β-MNTDC
  Arms: 11βmethyl nortestosterone dodecylcarbonate

SUMMARY:
The long term objective is to develop a new male hormone 11-β Methyl Nortestosterone Dodecylcarbonate (11β-MNTDC) as a male hormonal contraceptive.

DETAILED DESCRIPTION:
This is a Phase I multicenter, double-blind, single dose, dose-ranging study, in healthy men followed on an inpatient basis to evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics of 11β-methyl nortestosterone dodecylcarbonate (11β-MNTDC).

This single dose, dose-ranging study of 4 escalating doses will be conducted in two centers.

Initially, 12 men will be enrolled in total, 6 men at each center, with a goal of having a minimum of 12 healthy male subjects completing this study (10 active drugs and 2 placebos) both in the fed and fasting states at each dose.

Each of the 4 doses of 11β-MNTDC will be administered first fasting and then fed. Each of the doses of 11β-MNTDC will be administered about 28 days apart +/- 14 days with the time interval between the fasting and fed dosing will be approximately 7 days (-2/+9 days) and a 7 to 14 day washout will occur before dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of screening.
2. 18 to 50 years of age (inclusive).
3. BMI ≤ 33 calculated as weight in kg/ (height in m2).
4. No history of hormonal therapy use in the last three months prior to the first screening visit.
5. Subject agrees to use a recognized effective method of contraception with any female partner (i.e. at a minimum, use barrier plus and additional method of contraception) during the course of the study treatment and recovery phase.
6. Subjects will refrain from donating blood or plasma during the study period.
7. Subjects will be advised to refrain/abstain from alcoholic beverages and grapefruit juice during the study period.
8. Subjects will not use cannabis or any recreational drugs at least 2 weeks before completing screening and during the study.
9. In the opinion of the investigator, subject is able to comply with the protocol, understand and sign an informed consent and HIPAA form.
10. Does not meet any of the exclusion criteria.

Exclusion Criteria:

1. Men participating in another clinical trial involving an investigational drug within the last 30 days prior to the first screening visit.
2. Men not living in the catchment area of the clinic or within a reasonable distance from the study site.
3. Clinically significant abnormal physical and laboratory findings at screening.
4. Elevated PSA (levels ≥ 2.5 ng/mL), according to local laboratory normal values.
5. Abnormal serum chemistry values, according to local laboratory reference ranges that indicate liver or kidney dysfunction or that may be considered clinically significant except for: an upper limit for fasting bilirubin less than 2 mg/dL, upper limit for cholesterol less than 221 mg/dL, or upper limit for fasting triglycerides less than 201 mg/dL.
6. Use of androgens within 2 months before first screening visit.
7. Ongoing use of body building nutritional supplements.
8. Systolic BP > 135 mm Hg and Diastolic blood pressure BP > 85 and mm Hg; ((BP) Blood pressure will be taken 3 times at 5 - minute intervals and the mean of all measurements be considered).
9. Clinically significant abnormal EKG or a QTc interval of > 450 msec.
10. History of hypertension, including hypertension controlled with treatment.
11. Benign or malignant liver tumors; active liver disease.
12. History of breast carcinoma.
13. Known history of androgen deficiency due to hypothalamic-pituitary or testicular disease.
14. Known history of cardiovascular, renal, hepatic or prostatic disease or significant psychiatric illness.
15. Positive serology for active Hepatitis (not immunization-related serology) or HIV at screening visit.
16. A serious systemic disease such as diabetes mellitus or obesity (body weight greater than BMI >33 kg/m2 as above).
17. History of known, untreated sleep apnea.
18. Known or suspected alcoholism or drug abuse that may affect metabolism/transformation of steroid hormones or study treatment compliance.
19. Partner is known to be pregnant.
20. Men desiring fertility within the first 24 weeks of study participation.
21. Men participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine will be advised of the relative and temporary hazards that participating in this study may have for their sporting status.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single dose oral administration of up to 4 escalating doses of 11-β methyl nortestosterone dodecylcarbonate (11β-MNTDC) as measured by adverse events | 12-20 weeks
  As by adverse events
Safety and tolerability of single dose oral administration of up to 4 escalating doses of 11-β methyl nortestosterone dodecylcarbonate (11β-MNTDC) as measured by changes from baseline in vital signs | 12-20 weeks
  As by changes from baseline in vital signs
Safety and tolerability of single dose oral administration of up to 4 escalating doses of 11-β methyl nortestosterone dodecylcarbonate (11β-MNTDC) as measured by changes from baseline in electrocardiogram (EKG) | 12-20 weeks
  As by changes from baseline in EKG
Safety and tolerability of single dose oral administration of up to 4 escalating doses of 11-β methyl nortestosterone dodecylcarbonate (11β-MNTDC) as measured by changes from baseline in physical exams | 12-20 weeks
  As by changes from baseline in physical exams
Safety and tolerability of single dose oral administration of up to 4 escalating doses of 11-β methyl nortestosterone dodecylcarbonate (11β-MNTDC) as measured by changes from baseline in lab tests | 12-20 weeks
  As by changes from baseline in lab tests

SECONDARY OUTCOMES:
Pharmacokinetics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose using area under the curve (AUC) | 112 days
  11β-MNTDC PK levels at various time points through the 112 days of treatment using AUC
Pharmacokinetics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose using maximum concentration (Cmax) | 112 days
  11β-MNTDC PK levels at various time points through the 112 days of treatment using Cmax
Pharmacokinetics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose using Time to Reach Maximum Concentration (Tmax) | 112 days
  11β-MNTDC PK levels at various time points through the 112 days of treatment using Tmax
Pharmacodynamics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose as measured by Luteinizing Hormone (LH) | 112 days
  11β-MNTDC PD levels at various time points through the 112 days of treatment
Pharmacodynamics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose as measured by Follicle Stimulating Hormone (FSH) | 112 days
  11β-MNTDC PD levels at various time points through the 112 days of treatment
Pharmacodynamics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose as measured by Testosterone (T) | 112 days
  11β-MNTDC PD levels at various time points through the 112 days of treatment
Pharmacodynamics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose as measured by free Testosterone (free T) | 112 days
  11β-MNTDC PD levels at various time points through the 112 days of treatment
Pharmacodynamics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose as measured by Dihydrotestosterone (DHT) | 112 days
  11β-MNTDC PD levels at various time points through the 112 days of treatment
Pharmacodynamics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose as measured by estradiol (E2) | 112 days
  11β-MNTDC PD levels at various time points through the 112 days of treatment
Pharmacodynamics of 11β-MNTDC after 4 escalating oral doses of 11β-MNTDC administered in a fast and fed cycle lasting approximately 28 days for each dose as measured by Sex Hormone Binding Globulin (SHBG) | 112 days
  11β-MNTDC PD levels at various time points through the 112 days of treatment
Effect of food on the pharmacokinetics of orally administered 11β-MNTDC using Average Concentration (Cavg) | 112 days
  Comparison of pharmacokinetic measures among the single dose periods and comparison of PK parameters in the fed and fasting states will be performed with mixed model repeated measures analysis of variance (ANOVA). Evidence of lack of food effect will be concluded if ANOVA-estimated PK parameters (Cavg) after food are within 80 to 125% of those obtained at the fasting state.
Effect of food on the pharmacokinetics of orally administered 11β-MNTDC using the area under the curve from 0-24 hours (AUC 0-24h) | 112 days
  Comparison of pharmacokinetic measures among the single dose periods and comparison of PK parameters in the fed and fasting states will be performed with mixed model repeated measures analysis of variance (ANOVA). Evidence of lack of food effect will be concluded if ANOVA-estimated PK parameters (AUC0-24h) after food are within 80 to 125% of those obtained at the fasting state.
Effect of food on the pharmacokinetics of orally administered 11β-MNTDC using maximum concentration (Cmax) | 112 days
  Comparison of pharmacokinetic measures among the single dose periods and comparison of PK parameters in the fed and fasting states will be performed with mixed model repeated measures analysis of variance (ANOVA). Evidence of lack of food effect will be concluded if ANOVA-estimated PK parameters (Cmax) after food are within 80 to 125% of those obtained at the fasting state.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wang, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center; Stephanie Page, MD, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Amory JK, Anawalt BD, Bremner WJ, Matsumoto AM. Daily testosterone and gonadotropin levels are similar in azoospermic and nonazoospermic normal men administered weekly testosterone: implications for male contraceptive development. J Androl. 2001 Nov-Dec;22(6):1053-60. doi: 10.1002/j.1939-4640.2001.tb03445.x. PMID 11700852
- [Background] Amory JK, Bremner WJ. Oral testosterone in oil plus dutasteride in men: a pharmacokinetic study. J Clin Endocrinol Metab. 2005 May;90(5):2610-7. doi: 10.1210/jc.2004-1221. Epub 2005 Feb 15. PMID 15713724
- [Background] Anderson RA, Wallace AM, Wu FC. Comparison between testosterone enanthate-induced azoospermia and oligozoospermia in a male contraceptive study. III. Higher 5 alpha-reductase activity in oligozoospermic men administered supraphysiological doses of testosterone. J Clin Endocrinol Metab. 1996 Mar;81(3):902-8. doi: 10.1210/jcem.81.3.8772548.
- [Background] Attardi BJ, Engbring JA, Gropp D, Hild SA. Development of dimethandrolone 17beta-undecanoate (DMAU) as an oral male hormonal contraceptive: induction of infertility and recovery of fertility in adult male rabbits. J Androl. 2011 Sep-Oct;32(5):530-40. doi: 10.2164/jandrol.110.011817. Epub 2010 Dec 16. PMID 21164142
- [Background] Attardi BJ, Hild SA, Koduri S, Pham T, Pessaint L, Engbring J, Till B, Gropp D, Semon A, Reel JR. The potent synthetic androgens, dimethandrolone (7alpha,11beta-dimethyl-19-nortestosterone) and 11beta-methyl-19-nortestosterone, do not require 5alpha-reduction to exert their maximal androgenic effects. J Steroid Biochem Mol Biol. 2010 Oct;122(4):212-8. doi: 10.1016/j.jsbmb.2010.06.009. Epub 2010 Jun 25. PMID 20599615
- [Background] Attardi BJ, Hild SA, Reel JR. Dimethandrolone undecanoate: a new potent orally active androgen with progestational activity. Endocrinology. 2006 Jun;147(6):3016-26. doi: 10.1210/en.2005-1524. Epub 2006 Feb 23. PMID 16497801
- [Background] Attardi BJ, Marck BT, Matsumoto AM, Koduri S, Hild SA. Long-term effects of dimethandrolone 17beta-undecanoate and 11beta-methyl-19-nortestosterone 17beta-dodecylcarbonate on body composition, bone mineral density, serum gonadotropins, and androgenic/anabolic activity in castrated male rats. J Androl. 2011 Mar-Apr;32(2):183-92. doi: 10.2164/jandrol.110.010371. Epub 2010 Aug 26. PMID 20798389
- [Background] Attardi BJ, Pham TC, Radler LC, Burgenson J, Hild SA, Reel JR. Dimethandrolone (7alpha,11beta-dimethyl-19-nortestosterone) and 11beta-methyl-19-nortestosterone are not converted to aromatic A-ring products in the presence of recombinant human aromatase. J Steroid Biochem Mol Biol. 2008 Jun;110(3-5):214-22. doi: 10.1016/j.jsbmb.2007.11.009. PMID 18555683
- [Background] Bagchus WM, Hust R, Maris F, Schnabel PG, Houwing NS. Important effect of food on the bioavailability of oral testosterone undecanoate. Pharmacotherapy. 2003 Mar;23(3):319-25. doi: 10.1592/phco.23.3.319.32104. PMID 12627930
- [Background] Behre H M, Wang C, Handelsman D J & Nieschlag E. (2004) Pharmacology of Testosterone Preparations. In: Testosterone, Vol. Third (eds E Nieschlag & H M Behre), pp. 405-444. Cambridge University Press, Cambridge.
- [Background] Cook CE, Kepler JA. 7alpha,11beta-Dimethyl-19-nortestosterone: a potent and selective androgen response modulator with prostate-sparing properties. Bioorg Med Chem Lett. 2005 Feb 15;15(4):1213-6. doi: 10.1016/j.bmcl.2004.11.076. PMID 15686944
- [Background] Friedl KE, Hannan CJ Jr, Jones RE, Plymate SR. High-density lipoprotein cholesterol is not decreased if an aromatizable androgen is administered. Metabolism. 1990 Jan;39(1):69-74. doi: 10.1016/0026-0495(90)90150-b. PMID 2294373
- [Background] Gooren LJ. A ten-year safety study of the oral androgen testosterone undecanoate. J Androl. 1994 May-Jun;15(3):212-5. PMID 7928661
- [Background] Gu Y, Liang X, Wu W, Liu M, Song S, Cheng L, Bo L, Xiong C, Wang X, Liu X, Peng L, Yao K. Multicenter contraceptive efficacy trial of injectable testosterone undecanoate in Chinese men. J Clin Endocrinol Metab. 2009 Jun;94(6):1910-5. doi: 10.1210/jc.2008-1846. Epub 2009 Mar 17. PMID 19293262
- [Background] Heckel M J. (1939) Production of oliogspermia in a man by the use of testosterone propionate. Exl. Biol. Med. 40, 658-659.
- [Background] Hild SA, Attardi BJ, Koduri S, Till BA, Reel JR. Effects of synthetic androgens on liver function using the rabbit as a model. J Androl. 2010 Sep-Oct;31(5):472-81. doi: 10.2164/jandrol.109.009365. Epub 2010 Apr 8. PMID 20378929
- [Background] Houwing NS, Maris F, Schnabel PG, Bagchus WM. Pharmacokinetic study in women of three different doses of a new formulation of oral testosterone undecanoate, Andriol Testocaps. Pharmacotherapy. 2003 Oct;23(10):1257-65. doi: 10.1592/phco.23.12.1257.32707. PMID 14594344
- [Background] McLachlan RI, Robertson DM, Pruysers E, Ugoni A, Matsumoto AM, Anawalt BD, Bremner WJ, Meriggiola C. Relationship between serum gonadotropins and spermatogenic suppression in men undergoing steroidal contraceptive treatment. J Clin Endocrinol Metab. 2004 Jan;89(1):142-9. doi: 10.1210/jc.2003-030616. PMID 14715841
- [Background] Nieschlag E, Mauss J, Coert A, Kicovic P. Plasma androgen levels in men after oral administration of testosterone or testosterone undecanoate. Acta Endocrinol (Copenh). 1975 Jun;79(2):366-74. doi: 10.1530/acta.0.0790366. PMID 1173495
- [Background] Piotrowska K, Wang C, Swerdloff RS, Liu PY. Male hormonal contraception: hope and promise. Lancet Diabetes Endocrinol. 2017 Mar;5(3):214-223. doi: 10.1016/S2213-8587(16)00034-6. Epub 2016 Feb 23. PMID 26915313
- [Background] Qoubaitary A, Swerdloff RS, Wang C. Advances in male hormone substitution therapy. Expert Opin Pharmacother. 2005 Aug;6(9):1493-506. doi: 10.1517/14656566.6.9.1493. PMID 16086637
- [Background] Roth MY, Page ST, Bremner WJ. Male hormonal contraception: looking back and moving forward. Andrology. 2016 Jan;4(1):4-12. doi: 10.1111/andr.12110. Epub 2015 Oct 9. PMID 26453296
- [Background] Rothman MS, Carlson NE, Xu M, Wang C, Swerdloff R, Lee P, Goh VH, Ridgway EC, Wierman ME. Reexamination of testosterone, dihydrotestosterone, estradiol and estrone levels across the menstrual cycle and in postmenopausal women measured by liquid chromatography-tandem mass spectrometry. Steroids. 2011 Jan;76(1-2):177-82. doi: 10.1016/j.steroids.2010.10.010. Epub 2010 Nov 9. PMID 21070796
- [Background] Skakkebaek NE, Bancroft J, Davidson DW, Warner P. Androgen replacement with oral testosterone undecanoate in hypogonadal men: a double blind controlled study. Clin Endocrinol (Oxf). 1981 Jan;14(1):49-61. doi: 10.1111/j.1365-2265.1981.tb00364.x. PMID 7014044
- [Background] Surampudi P, Page ST, Swerdloff RS, Nya-Ngatchou JJ, Liu PY, Amory JK, Leung A, Hull L, Blithe DL, Woo J, Bremner WJ, Wang C. Single, escalating dose pharmacokinetics, safety and food effects of a new oral androgen dimethandrolone undecanoate in man: a prototype oral male hormonal contraceptive. Andrology. 2014 Jul;2(4):579-587. doi: 10.1111/j.2047-2927.2014.00216.x. Epub 2014 May 2. PMID 24789057
- [Background] Swerdloff RS, Wang C, Cunningham G, Dobs A, Iranmanesh A, Matsumoto AM, Snyder PJ, Weber T, Longstreth J, Berman N. Long-term pharmacokinetics of transdermal testosterone gel in hypogonadal men. J Clin Endocrinol Metab. 2000 Dec;85(12):4500-10. doi: 10.1210/jcem.85.12.7045. PMID 11134099
- [Background] Vermeulen A, Verdonck L, Kaufman JM. A critical evaluation of simple methods for the estimation of free testosterone in serum. J Clin Endocrinol Metab. 1999 Oct;84(10):3666-72. doi: 10.1210/jcem.84.10.6079. PMID 10523012
- [Background] von Eckardstein S, Noe G, Brache V, Nieschlag E, Croxatto H, Alvarez F, Moo-Young A, Sivin I, Kumar N, Small M, Sundaram K; International Committee for Contraception Research, The Population Council. A clinical trial of 7 alpha-methyl-19-nortestosterone implants for possible use as a long-acting contraceptive for men. J Clin Endocrinol Metab. 2003 Nov;88(11):5232-9. doi: 10.1210/jc.2002-022043. PMID 14602755
- [Background] Wang C, Catlin DH, Demers LM, Starcevic B, Swerdloff RS. Measurement of total serum testosterone in adult men: comparison of current laboratory methods versus liquid chromatography-tandem mass spectrometry. J Clin Endocrinol Metab. 2004 Feb;89(2):534-43. doi: 10.1210/jc.2003-031287. PMID 14764758
- [Background] Wang C, Shiraishi S, Leung A, Baravarian S, Hull L, Goh V, Lee PW, Swerdloff RS. Validation of a testosterone and dihydrotestosterone liquid chromatography tandem mass spectrometry assay: Interference and comparison with established methods. Steroids. 2008 Dec 12;73(13):1345-52. doi: 10.1016/j.steroids.2008.05.004. Epub 2008 May 21. PMID 18579171
- [Background] Wang C, Swerdloff R, Kipnes M, Matsumoto AM, Dobs AS, Cunningham G, Katznelson L, Weber TJ, Friedman TC, Snyder P, Levine HL. New testosterone buccal system (Striant) delivers physiological testosterone levels: pharmacokinetics study in hypogonadal men. J Clin Endocrinol Metab. 2004 Aug;89(8):3821-9. doi: 10.1210/jc.2003-031866. PMID 15292312
- [Background] Contraceptive efficacy of testosterone-induced azoospermia in normal men. World Health Organization Task Force on methods for the regulation of male fertility. Lancet. 1990 Oct 20;336(8721):955-9. PMID 1977002
- [Background] World Health Organization Task Force on Methods for the Regulation of Male Fertility. Contraceptive efficacy of testosterone-induced azoospermia and oligozoospermia in normal men. Fertil Steril. 1996 Apr;65(4):821-9. PMID 8654646
- [Derived] Yuen F, Thirumalai A, Fernando FA, Swerdloff RS, Liu PY, Pak Y, Hull L, Bross R, Blithe DL, Long JE, Page ST, Wang C. Comparison of metabolic effects of the progestational androgens dimethandrolone undecanoate and 11beta-MNTDC in healthy men. Andrology. 2021 Sep;9(5):1526-1539. doi: 10.1111/andr.13025. Epub 2021 May 22. PMID 33908182
- [Derived] Yuen F, Thirumalai A, Pham C, Swerdloff RS, Anawalt BD, Liu PY, Amory JK, Bremner WJ, Dart C, Wu H, Hull L, Blithe DL, Long J, Wang C, Page ST. Daily Oral Administration of the Novel Androgen 11beta-MNTDC Markedly Suppresses Serum Gonadotropins in Healthy Men. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e835-47. doi: 10.1210/clinem/dgaa032. PMID 31976519
- [Derived] Wu S, Yuen F, Swerdloff RS, Pak Y, Thirumalai A, Liu PY, Amory JK, Bai F, Hull L, Blithe DL, Anawalt BD, Parman T, Kim K, Lee MS, Bremner WJ, Page ST, Wang C. Safety and Pharmacokinetics of Single-Dose Novel Oral Androgen 11beta-Methyl-19-Nortestosterone-17beta-Dodecylcarbonate in Men. J Clin Endocrinol Metab. 2019 Mar 1;104(3):629-638. doi: 10.1210/jc.2018-01528. PMID 30252057